CLINICAL TRIAL: NCT01732718
Title: The Effect of Atorvastatin on Endothelial Dysfunction and Albuminuria in Sickle Cell Disease (in the Grant Entitled: Endothelial Dysfunction in the Pathogenesis of Sickle Cell Nephropathy)
Brief Title: Effect of Atorvastatin on Endothelial Dysfunction and Albuminuria in Sickle Cell Disease
Acronym: ENDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-1354; R01HL111659 (NIH)
Record Dates: First submitted 2012-11-09; First posted 2012-11-26 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2018-11

CONDITIONS: Sickle Cell Disease; Sickle Cell Nephropathy
Keywords: sickle cell disease; endothelial function; albuminuria; atorvastatin; soluble fms-like tyrosine kinase-1
MeSH Terms: conditions — Anemia, Sickle Cell; Albuminuria | interventions — Atorvastatin; Sugars; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin, then Placebo (Experimental): Participants first received Atorvastatin 40 mg tablets once daily for 6 weeks. After a washout period of 4 weeks, they then received placebo (matching Atorvastatin 40 mg tablets) once daily for 6 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo
- Placebo, Then Atorvastatin (Placebo Comparator): Participants first received Placebo (matching Atorvastatin 40 mg tablets) once daily for 6 weeks. After a washout period of 4 weeks, they then received Atorvastatin 40 mg tablets once daily for 6 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 40 mg tablet by mouth daily for 6 weeks
  Other Names: Lipitor®
Drug: Placebo — Matching placebo tablet by mouth daily for 6 weeks
  Other Names: Sugar pill manufactured to mimic atorvastatin 40 mg tablet

SUMMARY:
The purpose of this research study is to learn about the effect of the drug, atorvastatin, on blood vessels in patients with sickle cell disease.

The primary hypothesis is that endothelial dysfunction is an important contributor to the pathophysiology of albuminuria in SCD. The investigators propose that atorvastatin will improve endothelial dysfunction, decrease levels of soluble fms-like tyrosine kinase-1 (sFLT-1), and decrease albuminuria in SCD patients.

Participants will be individuals with sickle cell disease, age 18 to 60, who have some degree of albuminuria. A total of 19 subjects, males and females, will be enrolled. The study is made up of Screening, Treatment, and Follow Up phases and has a cross-over design. After patients are screened for eligibility, they will be randomized to receive atorvastatin or placebo in the initial six-week treatment period. When that is complete, there will be a four-week washout period before they begin another six-week treatment period. In the second treatment period, they "cross-over" to the other treatment arm. Four weeks after the end of the second treatment period, follow-up safety assessments will be done.

DETAILED DESCRIPTION:
It is well recognized that sickle cell disease (SCD) is characterized by a vasculopathy, with involvement of multiple organs including the brain, lung, spleen, and kidney. This results in multiple clinical complications, including ischemic stroke, pulmonary hypertension, autosplenectomy, as well as albuminuria and chronic renal disease. Several recent studies have confirmed the association of both albuminuria and renal dysfunction with echocardiographically-defined pulmonary hypertension and other vasculopathic complications in SCD, suggesting that they may share a similar pathophysiology. Despite the high prevalence of albuminuria in patients with SCD and the known association of renal failure with increased mortality, the pathophysiology and treatment of albuminuria in this setting remain poorly defined.

The treatment options for nephropathy in SCD are limited. Although Angiotensin converting enzyme (ACE) inhibitors are the "standard of care" in the treatment of patients with proteinuria, there are to date no controlled, long-term studies confirming their efficacy and safety in this setting.

In this study, the investigators will evaluate the efficacy and safety of atorvastatin in SCD patients. At the completion of this trial, the investigators will have an improved understanding of the contribution of endothelial dysfunction to the pathophysiology of albuminuria in SCD. If the data support the hypothesis that atorvastatin is safe and effective in this population, the investigators plan on carrying out adequately powered studies to more definitively evaluate its safety and efficacy in the treatment and/or prevention of albuminuria in SCD.

ELIGIBILITY:
Inclusion Criteria:

1. Sickle cell anemia (HbSS) or Sickle-beta0 thalassemia (HbS-beta0thal) between ages of 18 and 60;
2. albuminuria (micro- or macroalbuminuria, defined as =/> 30mg/g creatinine);
3. serum alanine aminotransferase (ALT) </= 2 times upper limits of normal and/or gamma-glutamyl transferase (GGT) </= 3 times upper limits of normal;
4. platelet count > 150,000 cu/mm;
5. normal baseline coagulation profile (PT, International Normalized Ratio (INR), and PTT);
6. non-crisis, steady state with no severe pain episodes during the preceding 4 weeks, and no documented infection in the 2 weeks prior to enrollment;
7. ability to understand the requirements of the study;
8. if a woman of childbearing potential, must use an adequate method of contraception; and
9. if receiving hydroxyurea, ACE inhibitors or angiotensin blockers (ARB), should be on a stable dose for at least 3 months.

Exclusion Criteria:

1. hypersensitivity to any component of atorvastatin, or history of adverse reaction to statins;
2. pregnant or breastfeeding;
3. on statin therapy;
4. history of metastatic cancer;
5. current history of alcohol abuse;
6. history of diabetes mellitus or poorly controlled systemic hypertension;
7. end-stage renal disease;
8. total cholesterol level < 80 mg/dL and LDL cholesterol > 130 mg/dL;
9. on a chronic transfusion program;
10. ingested any investigational drugs within the past 4 weeks;
11. prior history of any myopathy;
12. allergy to nitroglycerin;
13. taking any of the following drugs: phosphodiesterase-5 inhibitors (e.g., sildenafil), cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors (e.g., cyclosporine, protease inhibitors), macrolide antibiotics (e.g., clarithromycin, erythromycin), fibric acid derivatives (e.g. gemfibrozil), niacin, colchicines, antifungal agents (azole derivatives), amiodarone, danazol, daptomycin, diltiazem, verapamil, eltrombopag, everolimus, fosphenytoin, or lanthanum.

Patients will also be encouraged to avoid grape fruit juice and red yeast rice for the duration of the study.

Atorvastatin is contraindicated during pregnancy and breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MBBS, Principal Investigator — University of North Caroina at Chapel Hill
Locations (1):
- UNC School of Medicine Clinical&Translational Research Ctr, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Atorvastatin, Then Placebo | Placebo, Then Atorvastatin
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Atorvastatin, Then Placebo | Placebo, Then Atorvastatin
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Atorvastatin, Then Placebo | Placebo, Then Atorvastatin
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Atorvastatin 40 mg or Placebo (matching Atorvastatin 40 mg)
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [44 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Endothelial Function
Description: Endothelial function will be assessed using ultrasound imaging of the brachial artery, with measurement of endothelium-dependent (flow-mediated) and endothelium-independent (nitroglycerin-mediated) dilation of the artery measured in millimeters (mm).
Time Frame: Baseline, 6 weeks
Measure: Median (Inter-Quartile Range); unit: % diameter change
Groups:
- Atorvastatin: Participants who received Atorvastatin 40 mg tablet in either the first or the second intervention
- Placebo: Participants who received placebo tablet (matching Atorvastatin 40 mg) in either the first or the second intervention
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 13
% diameter change | 1.44 [-2.66 to 4.43] | 0.69 [-1.94 to 3.18]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority; p = 0.51, Student t-test followed by ANOVA; Student t-test subsequently followed by crossover ANOVA model testing carry-over effect and treatment effect

2. Secondary Outcome: Change From Baseline to Week 6 in Plasma Markers of Endothelial Activation
Description: Investigators will measure plasma levels of soluble vascular cell adhesion molecules (sVCAM) and soluble intracellular adhesion molecule (sICAM) at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Population: Investigators elected to look at only one marker of vascular endothelial injury, i.e. sVCAM, so there is no data for sICAM.
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 13
ng/mL | 22.99 [-58.8 to 41.7] | 7.54 [-75.2 to 149.9]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline to Week 6 in Heme Oxygenase Activity
Description: The expression and activity of heme oxygenase-1(HO-1)will be determined at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Population: Data not collected
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline to Week 6 in Plasma Levels of Soluble Fms-like Tyrosine Kinase-1 (sFLT-1)
Description: Investigators will measure plasma levels of soluble fms-like tyrosine kinase-1 (sFLT-1) at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 13
pg/mL | 19.2 [-47.1 to 47.7] | 36.9 [-20.9 to 129.6]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline to Week 6 in Monocyte Activation
Description: Flow cytometry performed to assess monocyte activation at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Population: The stored samples did not survive the freeze/thaw process and as such, this data was not attainable.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline to Week 6 in Renal Function
Description: Investigators will assess the effect of atorvastatin on albuminuria by spot urine microalbuminuria/creatinine ratio measured at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Measure: Median (Inter-Quartile Range); unit: ug per mg
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 13
ug per mg | 28.8 [-28.6 to 237.1] | 74.9 [-15.2 to 373.4]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority; p = 0.57, see comments for explanation; albuminuria examined as continuous variable (linear mixed model to analyze effect) and categorical generalized variable (estimating equation approach)

7. Secondary Outcome: Occurrence of Adverse Events.
Description: Subjects will be evaluated for safety by patient self-report of adverse events and results of laboratory tests.
Time Frame: Continuously from randomization through end of study
Measure: Number; unit: events
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 13
events | 9 | 13

8. Secondary Outcome: Abnormal Physical Findings.
Description: Subjects will be evaluated by physical examination and/or measurement of vital signs at each study visit.
Time Frame: Baseline, 2, 4, and 6 weeks during treatment, and at follow-up.
Measure: Number; unit: participants
Groups:
- Baseline-Atorvastatin; Week 4-Atorvastatin; Week 6-Atorvastatin: Participants receiving Atorvastatin 40 mg tablets once daily for 6 weeks
- Baseline-Placebo; Week 4-Placebo; Week 6-Placebo: Participants receiving Placebo once daily for 6 weeks
Arm/Group | Baseline-Atorvastatin | Week 4-Atorvastatin | Week 6-Atorvastatin | Baseline-Placebo | Week 4-Placebo | Week 6-Placebo
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13 | 13
participants | 0 | 2 | 1 | 1 | 0 | 1

9. Secondary Outcome: Change From Baseline to Week 6 in Rho/Rho Kinase Activity
Description: The expression and activity of rho/rho kinase will be determined at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Population: Due to loss of key study personnel these data were not collected
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline to Week 6 in Plasma Levels of Vascular Endothelial Growth Factor (VEGF)
Description: Investigators will measure plasma levels of vascular endothelial growth factor (VEGF) at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Measure: Mean (Inter-Quartile Range); unit: pg/mL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 13
pg/mL | -3.99 [-29.4 to 7.8] | -10.5 [-50.4 to 9.8]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Mean Change From Baseline to Week 6 in Absolute Cell Counts
Description: Flow cytometry will be performed to assess absolute cell counts at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Population: Intent was to perform analysis using flow cytometry but cells did not survive thawing. Decision was made to use CBC laboratory values for absolute monocyte (AMC), lymphocyte (ALC) and neutrophil (ANC) counts to perform the analysis.
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 12
10^9 cells/L
  AMC | -0.07 [-0.26 to 0.12] | 0.15 [-0.11 to 0.41]
  ALC | 0.08 [-0.34 to 0.49] | -0.22 [-0.85 to 0.42]
  ANC | -0.18 [-0.96 to 0.61] | -0.55 [-1.91 to 0.81]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Comparison of the change in AMC; Test type: Superiority; p = 0.1469, t-test, 1 sided
Statistical Analysis 2: Comparison: Atorvastatin vs Placebo; Comparison of the change in ALC; Test type: Superiority; p = 0.2382, t-test, 1 sided
Statistical Analysis 3: Comparison: Atorvastatin vs Placebo; Comparison of the change in ANC; Test type: Superiority; p = 0.5833, t-test, 1 sided

12. Secondary Outcome: Change From Baseline to Week 6 in Tissue Factor (TF) Expression
Description: Flow cytometry will be performed to assess TF expression at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Population: The stored samples did not survive the freeze/thaw process and as such, this data was not attainable.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline to Week 6 in TF-mediated sFLT Release From Monocytes
Description: Flow cytometry will be performed to assess TF-mediated sFLT release from monocytes at baseline and at 6 weeks of treatment.
Time Frame: Baseline, 6 weeks
Population: The stored samples did not survive the freeze/thaw process and as such, this data was not attainable.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline to Week 6 in Tricuspid Regurgitant (TR) Jet.
Description: Echocardiogram will be used to assess TR jet before and after treatment.
Time Frame: Baseline, Week 6
Measure: Mean (95% Confidence Interval); unit: m/sec
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 13 | 13
m/sec | 0.80 [-1.64 to 3.24] | -0.05 [-0.69 to 0.56]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; Test type: Superiority; p = 0.5184, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Beginning with the first intervention and throughout washout and second intervention and then for 4 weeks after end of treatment
Arm/Group | Atorvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13 | 3/13
Other Adverse Events (participants affected / at risk) | 7/13 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=13) | Placebo (N=13)
Pain Crisis (Vascular disorders) | 1 (1) | 3 (3)
Heart Palpitations and Fainting (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=13) | Placebo (N=13)
Influenza B (Infections and infestations) | 0 (0) | 1 (1)
Headaches/Head Pressure (General disorders) | 2 (3) | 0 (0)
Pain Crisis Treated at Home (Vascular disorders) | 1 (1) | 2 (2)
Dry Skin (General disorders) | 0 (0) | 2 (2)
Edema of Lower Extremity (Vascular disorders) | 1 (1) | 1 (1)
Leg Ulcer (Vascular disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Low O2 Saturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea and Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Low ANC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Axillary Adenopathy (General disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left Wrist Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was limited by its small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT01732718/Prot_SAP_000.pdf